CLINICAL TRIAL: NCT03458429
Title: Safety and Efficacy of GMFFP From Young Healthy Donors (18-35), Treated With G-CSF to Ameliorate Frailty and Enhance the Immune Risk Profile in Older Individuals
Brief Title: Safety, Efficacy of FFP From Healthy Donors to Ameliorate Frailty and Enhance Immune Function in Older Individuals
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dipnarine Maharaj (Other)
Responsible Party: Sponsor-Investigator, Dipnarine Maharaj, Principal Investigator, South Florida Bone Marrow/Stem Cell Transplant Institute
Organization: South Florida Bone Marrow/Stem Cell Transplant Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001.16-BMSCTI
Record Dates: First submitted 2018-02-07; First posted 2018-03-08 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Frailty
Keywords: Young Donor Plasma; Frailty; Aging; Immune Function; G-CSF
MeSH Terms: conditions — Frailty | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: To determine the safety and tolerability of 12 once monthly transfusions of GMFFP (Granulocyte - Colony Stimulating Factor (G-CSF) Mobilized Fresh Frozen Plasma harvested from young, healthy donors), given to older, frail individuals who are at risk due to unhealthy aging and who will then have a subsequent 12-month follow-up period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Frail, older subjects (Experimental): Treated subjects are the frail, older subjects who will be treated with Granulocyte-Colony Stimulating Factor (G-CSF) Mobilized Fresh Frozen Plasma (GMFFP) in this protocol.
  Interventions: Drug: GMFFP

INTERVENTIONS:
Drug: GMFFP — Granulocyte-Colony Stimulating Factor (G-CSF) Mobilized Fresh Frozen Plasma
  Other Names: Granulocyte-Colony Stimulating Factor (G-CSF) Young Plasma

SUMMARY:
1. Primary Objective

   To determine the safety and tolerability of 12 once monthly transfusions of GMFFP (Granulocyte - Colony Stimulating Factor (G-CSF) Mobilized Fresh Frozen Plasma harvested from young, healthy donors), given to older, frail individuals who are at risk due to unhealthy aging and who will then have a subsequent 12-month follow-up period.
2. Secondary Objective

To determine the efficacy in older, frail individuals of 12 once monthly transfusions of GMFFP (Granulocyte - Colony Stimulating Factor (G-CSF) Mobilized Fresh Frozen Plasma harvested from young, healthy donors), and a subsequent 12-month follow-up period, to improve the Immune Risk Profile, ("IRP"), cognitive function (MME), quality of life (OPQOL-35), Frailty Index ("FI"), associated with unhealthy aging in the treated subjects.

DETAILED DESCRIPTION:
There have been recent reports in medical literature about the discovery that young mice's blood plasma when infused into aged mice caused regeneration of organs such as liver, and brain. There are certain factors present in the young blood which have been shown to improve the function of the organs.

In humans, transferring of young blood plasma to treat the effect of aging has already been attempted by a few doctors. In addition, fresh frozen blood plasma is currently used to treat patients who have disorders of blood clotting and immune disorders and is regarded as the standard of care by the medical community and as a safe treatment.

Over the past 25 years, peripheral blood stem cells (PBSC) concentrates have replaced bone marrow as the source for autologous stem cell transplants. Each year approximately 20,000 healthy individuals receive a protein call Granulocyte Colony Stimulating Factor (G-CSF) in order to stimulate and release stem cells from the bone marrow into the peripheral blood and these stem cells are collected and reinfused into patients who have blood cancers and other immune disorders. Granulocyte Colony Stimulating Factor (G-CSF) has been approved by the FDA for mobilization of the stem cells and collection of an individual's own stem cells. In a standard peripheral blood stem cell transplant the stem cells as well as the plasma are collected from the donor and is reinfused into the patient for treatment. There are recent reports in the medical literature that mobilized stem cells secrete certain factors into the plasma of the blood and that these factors may be important for the regenerative capabilities of stem cells.

The transfusion of the plasma which contains these factors, secreted by the stem cells, which come from young individuals and are free of stem cells, may be an effective treatment for frailty and immune dysfunction in older individuals.

In this study, the treatment is considered experimental (investigational) because we are evaluating the safety and effectiveness of healthy donor plasma which contains the factors secreted by stem cells for the treatment of frailty and immune dysfunction. The plan of this study is to enroll about 30 subjects for treatment and follow up evaluation over a time period of two years (24 months).

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Be aged between 55-95 years.
* Show signs of frailty apart from a concomitant condition as assessed by the Investigator with a score of 4-7 on the Clinical Frailty Scale (Appendix 1) and/or Have an abnormal Immune Risk Profile (IRP)
* Not be pregnant or nursing while participating in this trial. Both men and women of reproductive potential must agree to use an effective means of birth control while participating in the trial. Women of childbearing potential should have a negative serum pregnancy test before treatment, if not surgically sterile.
* Have a negative neutrophil antibody test.
* Have a negative Human Leukocyte Antigen (HLA) Class I and II antibody test.
* Have Cytomegalovirus (CMV) negative or positive sero-testing completed.
* Have a life expectancy of at least 24 months as judged by the PI at the time of consent.
* Have less than 4 weeks since prior medical therapy, radiation therapy, and/or surgery
* Have adequate organ function including:

Hemoglobin greater than 10.0 g/dl Absolute neutrophils must be greater than 1,500/Microliter(uL) Platelet count must be greater than100,000/uL Serum bilirubin must be less than 2mg/dL Aspartate Aminotransferase (AST) must be less than 90 units/L Alanine Transaminase (ALT) must be less than 105 units/L Serum creatinine must be less than 2mg/dL

Exclusion Criteria:

* Have a score of less than 4 or greater than 7 on the Clinical Frailty Scale or Have a score of less than 4 and a No Immune Risk Profile (IRP)
* Have used anti-inflammatory medications within 7 days of study treatment,treated subjects may be re-screened after 14 days
* Abnormal clinical values including but not limited to:

Platelet count less than 100,000/mm3 Absolute neutrophils less than 1500/uL Hemoglobin less than 10 g/dL Aspartate transaminase, alanine transaminase, or alkaline phosphatase Greater than 3 times upper limit of normal Serum bilirubin greater than 2 mg/dL

* Be an organ transplant recipient or have an active listing (or expected future listing) for transplant of any organ.
* Have a documented intolerance to plasma or its components, or prior intolerance to intravenous fluids.
* Have known serum antibodies to plasma proteins, such as haptoglobin, Complement Component (C3/C4), or alpha-1-antitrypsin.
* Previous plasma transfusion within 30 days of signing informed consent.
* Serious comorbid illness including, but not limited to:

HIV or hepatitis Congenital deficiency of immunoglobulin A (IgA) Pulmonary edema Advanced liver or renal failure Uncontrolled diabetes mellitus, Significant and/or symptomatic cardiovascular disease (e.g. any history of myocardial infarction, congestive heart failure, unstable angina, uncontrolled arrhythmia) Active serious infection. Hemorrhagic cystitis Cardiac revascularization within last six months Severe obstructive ventilatory defect Renal insufficiency (serum creatinine greater than 177 mol/L or creatinine clearance less than 20 mL/min) Sickle cell disease or hemoglobinopathy Cancer Any other condition that the investigator believes may compromise the safety or compliance of the patient or the study evaluation.

* No vascular access
* Pregnant or nursing female
* Recent ( less than 24 months) history of drug or alcohol abuse
* Current participation in an investigational therapeutic or medical device trial
* Treatment with any human blood product, including intravenous immunoglobulin, during the 6 months prior to screening or during the trial.
* Recent use (within 30 days) of immunosuppressive agents
* Inability to perform any assessments or relevant procedures required for the study or to give informed consent

Although not considered a part of the formal eligibility criteria, the treating physicians will evaluate additional factors that may increase subject risk, including but not limited to:

The presence of serious illnesses that would limit survival to less than two years.

The presence of psychiatric conditions that would prevent compliance with study visits or impact informed consent.

The presence of uncontrolled or severe cardiovascular disease, pulmonary disease, age-related or other serious medical conditions, or infection, which, in the opinion of the treating physician, would make study participation unreasonably hazardous.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by clinical symptoms, laboratory abnormalities, serious adverse events and treatment-limiting adverse events | 24 months
  To determine the safety and tolerability of 12 once monthly transfusions of GMFFP (Granulocyte - Colony Stimulating Factor (G-CSF) Mobilized Fresh Frozen Plasma harvested from young, healthy donors) given to older, frail individuals who are at risk due to unhealthy aging and who will be assessed throughout the duration of treatment. After the one-year treatment period, participants will complete follow-up assessments every 3 months for 1 year.

SECONDARY OUTCOMES:
Efficacy outcomes as measured by changes from baseline at 12 and 24 months assessing Immune Risk Profile (IRP) | 12 and 24 months
  To determine the efficacy in older, frail individuals of 12 once monthly transfusions of GMFFP (Granulocyte - Colony Stimulating Factor (G-CSF) Mobilized Fresh Frozen Plasma harvested from young, healthy donors), and a subsequent 12-month follow-up period, to improve the Immune Risk Profile (IRP) as assessed by aging, inflammation and immune function biomarkers.
Efficacy outcomes as measured by changes from baseline at 12 and 24 months assessing cognitive function (MME) | 12 and 24 months
  To determine the efficacy in older, frail individuals of 12 once monthly transfusions of GMFFP (Granulocyte - Colony Stimulating Factor (G-CSF) Mobilized Fresh Frozen Plasma harvested from young, healthy donors), and a subsequent 12-month follow-up period, to improve cognitive function (MME) as assessed by cognitive impairment and to follow the course of cognitive changes in an individual over time. The test examines functions, including registration, attention and calculation, recall, language, ability to follow simple commands, and orientation.
Efficacy outcomes as measured by changes from baseline at 12 and 24 months assessing quality of life (OPQOL-35) | 12 and 24 months
  To determine the efficacy in older, frail individuals of 12 once monthly transfusions of GMFFP (Granulocyte - Colony Stimulating Factor (G-CSF) Mobilized Fresh Frozen Plasma harvested from young, healthy donors), and a subsequent 12-month follow-up period, to improve quality of life (OPQOL-35) assessed by the effect of health, social relationships, independence, psychological well-being, and activities on overall quality of life in older individuals
Efficacy outcomes as measured by changes from baseline at 12 and 24 months assessing Frailty Index (FI) | 12 and 24 months
  To determine the efficacy in older, frail individuals of 12 once monthly transfusions of GMFFP (Granulocyte - Colony Stimulating Factor (G-CSF) Mobilized Fresh Frozen Plasma harvested from young, healthy donors), and a subsequent 12-month follow-up period, to improve Frailty Index ("FI"), as measured by eight frailty factors including nutritional status, physical activity, mobility, energy, strength, cognition, mood, and social support

CONTACTS AND LOCATIONS:
Overall Officials: Dipnarine Maharaj, Principal Investigator — South Florida Bone Marrow/Stem Cell Transplant Institute
Locations (1):
- South Florida Bone Marrow/Stem Cell Transplant Institute DBA Maharaj Institute of Immune Regenerative Medicine, Boynton Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No